CLINICAL TRIAL: NCT00003049
Title: A Prospective, Randomized Trial of Extended Lymphadenectomy in the Management of Resectable Pancreatic Cancer
Brief Title: Surgery Followed by Radiation Therapy and Chemotherapy in Treating Patients With Cancer of the Pancreas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Randall K. Pearson, M.D., Mayo Clinic Cancer Center
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065689; P30CA015083 (NIH); 974301 (Other: Mayo Clinic Cancer Center); G97-1302 (Other: NCI Protocol); 152-97 (Other: Mayo Clinic IRB)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2011-05

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Leucovorin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluorouracil
Drug: leucovorin calcium
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Surgery to remove the pancreas, some of the small intestine, and lymph nodes may be more effective treatment for cancer of the pancreas than surgery to remove the pancreas and some of the small intestine alone. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining surgery, radiation therapy, and chemotherapy may be an effective treatment for cancer of the pancreas.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery to remove the pancreas and a portion of the small intestine with or without removing lymph nodes, followed by radiation therapy and chemotherapy, in treating patients with cancer of the pancreas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the overall survival of patients with resectable ductal pancreatic adenocarcinoma undergoing extended versus standard pancreatoduodenectomy.

OUTLINE: Patients are randomized to undergo standard pancreatoduodenectomy (PD) or PD with extended lymph node resection after an exploratory laparotomy.

Patients receive adjuvant chemoradiation therapy 4-6 weeks after surgery, if no metastases are evident. Radiation therapy is given every week for 5 weeks. Fluorouracil/leucovorin calcium is administered by rapid IV push daily within 2 hours of radiation on days 1-4 of week 1 and days 29-31 of week 5.

Patients are followed every 4 months for the first year, then every 6 months for the next 2 years.

PROJECTED ACCRUAL: 50 patients will be accrued per group for a total of 100 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven adenocarcinoma of the exocrine pancreas excluding periampullary cancer
* Resectable malignancy must be located in a region that can be encompassed by a radiation port of 20 x 20 cm
* No evidence of extranodal metastatic disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Bilateral renal function as demonstrated by excretory urogram (IVP) or abdominal CT scan with contrast OR
* Greater than 2/3 of one functioning kidney must be shielded during radiation therapy

Other:

* Must have adequate oral nutrition (greater than 1200 calories daily)
* Greater than 5 years since prior malignancy except:

  * Squamous cell skin cancer
  * Basal cell skin cancer
  * In situ cervical cancer
* Not pregnant or lactating
* Patients of reproductive potential must use effective birth control
* No cystic neoplasms of the pancreas
* No islet cell, periampullary or cholangiocarcinoma
* No Federal Medical Center inmates

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for this disease

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiation therapy for this disease
* No prior radiation therapy to the abdomen

Surgery:

* Celiotomy and standardized exploration for resectability required

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 1997-05; Primary Completion 2005-08 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall K. Pearson, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States